CLINICAL TRIAL: NCT06929546
Title: Anti-phospholipid Antibodies in Adult Patients With Different Clinical Manifestations of Lyme Borreliosis
Brief Title: Anti-phospolipid Antibodies in Lyme Borreliosis
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Petra Bogovič, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 0120-571/2024-2711-3
Record Dates: First submitted 2025-04-04; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Patients With Different Manifestations of Lyme Borreliosis; Persons With Nonspecific Symptoms and Positive Borrelia Antibodies in Serum; Blood Donors
Keywords: Lyme borreliosis; Erythema migrans; Lyme neuroborreliosis; Lyme arthritis; Acrodermatitis chronica atrophicans; Anti-phospholipid antibodies
MeSH Terms: conditions — Lyme Disease; Glossitis, Benign Migratory; Lyme Neuroborreliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with different well-defined manifestations of Lyme borreliosis: 150 patients with well-defined Lyme borreliosis of which: 30 presented with solitary erythema migrans (EM), 30 with multiple EM (MEM), 30 with Lyme neuroborreliosis (LNB), 30 with Lyme arthritis (LA), 30 with acrodermatitis chronica atrophicans (ACA).
  Interventions: Diagnostic Test: Anti-phospholipid antibodies
- Patients with nonspecific symptoms and positive borrelial antibodies in serum.: 50 patients with nonspecific symptoms and positive borrelial antibodies in serum.
  Interventions: Diagnostic Test: Anti-phospholipid antibodies
- Blood donors: 40 healthy blood donors.
  Interventions: Diagnostic Test: Anti-phospholipid antibodies

INTERVENTIONS:
Diagnostic Test: Anti-phospholipid antibodies — Serum samples will be obtained for determination of IgG and IgM isotypes of 4 anti-phospholipid antibodies including anti-cardiolipin (aCL), anti-phosphatidylserine (aPS), anti-phosphatidic acid (aPA) and anti-phosphatidylcholine (aPC) with in-house ELISAs.

SUMMARY:
Background Lyme borreliosis, caused by Borrelia burgdorferi sensu lato is transmitted to humans through the bite of an infected Ixodes tick. B. burgdorferi sensu lato accumulates intact phospholipids from its environment to support its growth. Several of these environmentally acquired phospholipids including phosphatidylserine, phosphatidylcholine and phosphatidic acid may be recognized by anti-phospholipid antibodies that are believed to arose early in infection. Here we aimed to investigate the levels of anti-phospholipid antibodies in patients with Lyme borreliosis.

Methods

Participants included in the study:

* 150 patients with well-defined Lyme borreliosis, of which 30 presented with solitary erythema migrans (EM), 30 with multiple EM (MEM), 30 with Lyme neuroborreliosis (LNB), 30 with Lyme arthritis (LA), 30 with acrodermatitis chronica atrophicans (ACA);
* 50 patients with nonspecific symptoms and positive borrelial antibodies in serum; and
* 40 healthy blood donors (control group; samples from healthy blood donors were used to determine the threshold for the assays).

Specimens:

* 4 serum samples from each individual patient with well-defined Lyme borreliosis (1 before antibiotic treatment, 3 during follow-up up to 1 year);
* 2 serum samples from patients with nonspecific symptoms and positive borrelial antibodies (1 before antibiotic treatment and one 3 months later);
* healthy blood donors: 1 serum specimen.

Anti-phospolipid antibodies:

Levels of IgG and IgM isotypes of 4 anti-phospholipid antibodies including anti-cardiolipin (aCL), anti-phosphatidylserine (aPS), anti-phosphatidic acid (aPA) and anti-phosphatidylcholine (aPC) will be analyzed with in-house ELISAs.

ELIGIBILITY:
Inclusion Criteria:

Fulfillment of clinical case definition criteria for European Lyme borreliosis (doi: 10.1111/j.1469-0691.2010.03175.x.).

Exclusion Criteria:

Autoimmune diseases, acute myocardial infarction, acute deep vein thrombosis, pregnancy, syphilis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Adult patients diagnosed with well-defined manifestations of Lyme borreliosis (according to European case definition) at the Outpatient Lyme borreliosis clinic.
  2. Adult patients with nonspecific symptoms and positive borrelial antibodies in serum referred to Outpatient Lyme borreliosis clinic.
  3. Adult healthy blood donors.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Anti-phospholipid antibody levels in well-defined clinical manifestations of Lyme disease before antibiotic treatment. | Baseline
  In all patients with well-defined Lyme borreliosis (EM, multiple EM, LNB, LA, ACA) levels of anti-phospholipid antibodies (AUG/AUM) will be determined before antibiotic treatment.
Levels of anti-phospholipid antibodies in patients with well-defined Lyme borreliosis (EM, multiple EM, LNB, LA, ACA) during the 1-year follow-up after antibiotic treatment.herapy in patients with well-defined Lyme borreliosis | Up to one year.
  Antiphospholipid antibody levels (AUG/AUM) will be determined in 3 serum samples from each individual patient with well-defined Lyme borreliosis during follow-up up to 1 year.

SECONDARY OUTCOMES:
Levels of anti-phospholipid antibodies in patients with nonspecific symptoms and positive borrelial antibodies in serum. Levels of anti-phospholipid antibodies in control group (healthy blood donors). | 3 months
  Determination of anti-phospholipid antibodies (AUG/AUM) in patients with nonspecific symptoms and positive borrelial antibodies will be determined before antibiotic treatment and 3 months later.
  Determination of anti-phospholipid antibodies in healthy blood donors (one specimen per donor).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No